CLINICAL TRIAL: NCT06914219
Title: Implementing an Interdisciplinary Eating Disorder Screening and Treatment Program for Post-Bariatric Surgery Patients in Nova Scotia
Acronym: TEAM-ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aaron Keshen (Other)
Collaborators: Queen Elizabeth II Health Sciences Centre Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Aaron Keshen, Psychiatrist and Co-director of the Nova Scotia Provincial Service for Eating Disorders, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TEAM-ED
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Bariatric Surgery Patients; Disordered Eating Behaviors
MeSH Terms: conditions — Disordered Eating Behavior | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TEAM-ED Program (Experimental)
  Interventions: Behavioral: Treatment and Evaluation for After Metabolic Surgery with Eating Disorders (TEAM-ED) Program

INTERVENTIONS:
Behavioral: Treatment and Evaluation for After Metabolic Surgery with Eating Disorders (TEAM-ED) Program — A program that combines a) streamlined access to screening, diagnostic assessment, and treatment (brief cognitive behaviour therapy [CBT-T]), b) an interdisciplinary team approach to treatment planning, for managing disordered eating in patients post-weight loss surgery.

SUMMARY:
The goal of this interventional study is to evaluate the Treatment and Evaluation for After Metabolic Surgery with Eating Disorders (TEAM-ED) program, which combines streamlined access to screening, diagnostic assessment, and treatment with an interdisciplinary team approach to treatment planning, for managing disordered eating in adults who have recently had weight loss surgery in Nova Scotia. The main question it aims to answer is 'can an interdisciplinary program for identifying and managing disordered eating after weight loss surgery be implemented in Nova Scotia?

This study will determine the feasibility and impact of the TEAM-ED program by assessing the following objectives:

1. Reach (how effectively the program engages the target population [post-weight loss surgery patients])
2. Effectiveness (the extent of the program's impact on key clinical outcomes related to disordered eating and weight management)
3. Adoption (the extent to which the program is adopted and accepted by clinicians)
4. Implementation (how consistent program delivery is and factors impacting consistent delivery)

Participants will complete a disordered eating screening questionnaire online every 3 months after weight loss surgery until they reach 18-months post-surgery. Participants found to have disordered eating will be referred to the Nova Scotia Provincial Eating Disorder Service (NSEDPS) for standard disordered eating treatment (brief cognitive behavioral therapy [CBT-T]) plus treatment plan oversight by both weight loss surgery and eating disorder specialists. Standard outcome measures will be collected at baseline, during eating disorder treatment, post-treatment, and at follow-ups. Participants may also be asked to do a one-on-one research interview about their experiences with the program.

ELIGIBILITY:
Inclusion Criteria:

* ≥19 years old
* Between 3- and 18-months post-weight loss surgery.
* Able to complete English computer-based self-report questionnaires (with adequate accommodation, if necessary).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Screening Engagement Rate | From the post-weight loss surgery timepoint when a participant is first enrolled in the screening procedure (3-, 6-, 9-, 12-, 15-, or 18-months) until 18-months post-surgery or until they screen positive for disordered eating.
  Percentage of eligible patients (i.e., post-weight loss patients who are enrolled in the screening procedure) who complete the disordered eating screening measure (i.e., Loss of Control Over Eating Scale [LOCES]) at each timepoint (3-, 6-, 9-, 12-, 15-, and 18-month). To be calculated with the equation: [Actual # of LOCES completed at a timepoint] / [Total # of eligible patients who could have completed LOCES at that timepoint]

SECONDARY OUTCOMES:
Screening Initiation Rate | From 3- to 18-months post-weight loss surgery.
  Percentage of eligible patients (i.e., those who are 3- to 18-months post-weight loss surgery and receiving follow-up care at the study clinics) who initiate the screening procedure. This will be calculated using the equation: [number of patients who fill out their initial screening questionnaire] / [number of patients registered for follow-up care post-weight loss surgery at the study clinics]. *Screening questionnaire is the Loss of Control Over Eating Scale (LOCES).
Proportion of eligible patients who screen positive for loss of control eating. | From 3- to 18-months post-weight loss surgery.
  Proportion of eligible patients (i.e., those enrolled in the screening procedure) who are identified via screening questionnaire as having loss of control eating. This will be calculated using the equation: [number of patients who screen positive for loss of control eating] / [number of patients enrolled in screening procedure]. *Screening questionnaire is the Loss of Control Over Eating Scale (LOCES).
Proportion of eligible patients who undergo a disordered eating diagnostic interview. | From the post-weight loss surgery timepoint when a participant is first enrolled in the screening procedure (3-, 6-, 9-, 12-, 15-, or 18-months) until they screen positive for disordered eating.
  Proportion of eligible patients (i.e., those who screen positive for disordered eating) who complete a disordered eating diagnostic interview led by a clinician using the Eating Disorder Examination - Bariatric Surgery Version (EDE-BSV).
Proportion of eligible patients who are diagnosed with disordered eating. | From the post-weight loss surgery timepoint when a participant is first enrolled in the screening procedure (3-, 6-, 9-, 12-, 15-, or 18-months) until they screen positive for disordered eating.
  Proportion of eligible patients (i.e., those in the screening procedure who screen positive then attend a disordered eating diagnostic interview) who are diagnosed with disordered eating by the clinician conducting the interview based on the results of that assessment.
Proportion of eligible patients who start disordered eating treatment. | From the post-weight loss surgery timepoint when a participant is first enrolled in the screening procedure (3-, 6-, 9-, 12-, 15-, or 18-months) until they screen positive for disordered eating.
  Proportion of eligible patients (i.e., those diagnosed with disordered eating following diagnostic interview) who choose to start treatment for disordered eating.
Change in disordered eating symptom frequency from baseline to post-treatment. | From baseline to post-treatment (Week 10).
  Patients in TEAM-ED treatment will complete the Eating Disorder Examination Questionnaire (EDE-Q) before and after the core sessions of brief cognitive behavior therapy (i.e., Week 10).
Change in disordered eating psychopathology severity from baseline to Week 4. | From baseline to Week 4.
  Patients in TEAM-ED treatment will complete the Eating Disorder Examination Questionnaire (EDE-Q) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. EDE-Q global scores range from 0-6, with higher scores indicating increased severity of eating disorder psychopathology.
Change in disordered eating psychopathology severity from baseline to post-treatment (Week 10). | From baseline to post-treatment (Week 10).
  Patients in TEAM-ED treatment will complete the Eating Disorder Examination Questionnaire (EDE-Q) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. EDE-Q global scores range from 0-6, with higher scores indicating increased severity of eating disorder psychopathology.
Change in disordered eating psychopathology severity from baseline to 1-month follow-up. | From baseline to 1-month follow-up (i.e., 1 month after Week 10).
  Patients in TEAM-ED treatment will complete the Eating Disorder Examination Questionnaire (EDE-Q) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. EDE-Q global scores range from 0-6, with higher scores indicating increased severity of eating disorder psychopathology.
Change in disordered eating psychopathology severity from baseline to 3-month follow-up. | From baseline to 3-month follow-up (i.e., 3 months after Week 10).
  Patients in TEAM-ED treatment will complete the Eating Disorder Examination Questionnaire (EDE-Q) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. EDE-Q global scores range from 0-6, with higher scores indicating increased severity of eating disorder psychopathology.
Change in anxiety symptom severity from baseline to Week 4. | From baseline to Week 4.
  Patients in TEAM-ED treatment will complete the Generalized Anxiety Disorder Scale (GAD-7) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. GAD-7 total scores range from 0 to 21, with higher scores indicating greater severity of generalized anxiety symptoms.
Change in anxiety symptom severity from baseline to post-treatment (Week 10). | From baseline to post-treatment (Week 10).
  Patients in TEAM-ED treatment will complete the Generalized Anxiety Disorder Scale (GAD-7) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. GAD-7 total scores range from 0 to 21, with higher scores indicating greater severity of generalized anxiety symptoms.
Change in anxiety symptom severity from baseline to 1-month follow-up. | From baseline to 1-month follow-up (i.e., 1 month after Week 10).
  Patients in TEAM-ED treatment will complete the Generalized Anxiety Disorder Scale (GAD-7) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. GAD-7 total scores range from 0 to 21, with higher scores indicating greater severity of generalized anxiety symptoms.
Change in anxiety symptom severity from baseline to 3-month follow-up. | From baseline to 3-month follow-up (i.e., 3 months after Week 10).
  Patients in TEAM-ED treatment will complete the Generalized Anxiety Disorder Scale (GAD-7) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. GAD-7 total scores range from 0 to 21, with higher scores indicating greater severity of generalized anxiety symptoms.
Change in depression symptom severity from baseline to Week 4. | From baseline to Week 4.
  Patients in TEAM-ED treatment will complete the Patient Health Questionnaire (PHQ-9) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. PHQ-9 total scores range from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
Change in depression symptom severity from baseline to post-treatment (Week 10). | From baseline to post-treatment (Week 10).
  Patients in TEAM-ED treatment will complete the Patient Health Questionnaire (PHQ-9) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. PHQ-9 total scores range from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
Change in depression symptom severity from baseline to 1-month follow-up. | From baseline to 1-month follow-up (i.e., 1 month after Week 10).
  Patients in TEAM-ED treatment will complete the Patient Health Questionnaire (PHQ-9) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. PHQ-9 total scores range from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
Change in depression symptom severity from baseline to 3-month follow-up. | From baseline to 3-month follow-up (i.e., 3 months after Week 10).
  Patients in TEAM-ED treatment will complete the Patient Health Questionnaire (PHQ-9) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. PHQ-9 total scores range from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
Change in psychosocial impairment from baseline to Week 4. | From baseline to Week 4.
  Patients in TEAM-ED treatment will complete the Clinical Impairment Assessment (CIA) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. CIA total scores range from 0 to 48, with higher scores indicating greater psychosocial impairment due to eating disorder symptoms.
Change in psychosocial impairment from baseline to post-treatment (Week 10). | From baseline to post-treatment (Week 10).
  Patients in TEAM-ED treatment will complete the Clinical Impairment Assessment (CIA) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. CIA total scores range from 0 to 48, higher scores indicating greater psychosocial impairment due to eating disorder symptoms.
Change in psychosocial impairment from baseline to 1-month follow-up. | From baseline to 1-month follow-up (i.e., 1 month after Week 10).
  Patients in TEAM-ED treatment will complete the Clinical Impairment Assessment (CIA) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. CIA total scores range from 0 to 48, higher scores indicating greater psychosocial impairment due to eating disorder symptoms.
Change in psychosocial impairment from baseline to 3-month follow-up. | From baseline to 3-month follow-up (i.e., 3 months after Week 10).
  Patients in TEAM-ED treatment will complete the Clinical Impairment Assessment (CIA) at baseline, Week 4, post-treatment (Week 10), 1-month follow-up, and 3-month follow-up. CIA total scores range from 0 to 48, higher scores indicating greater psychosocial impairment due to eating disorder symptoms.
Change in weight from baseline to Week 4. | From baseline to Week 4.
  Patient weight as measured with a standard scale.
Change in weight from baseline to post-treatment (Week 10). | From baseline to post-treatment (Week 10).
  Patient weight as measured with a standard scale.
Change in weight from baseline to 1-month follow-up. | From baseline to 1-month follow-up (i.e., 1 month after Week 10).
  Patient weight as measured with a standard scale.
Change in weight from baseline to 3-month follow-up. | From baseline to 3-month follow-up (i.e., 3 months after Week 10).
  Patient weight as measured with a standard scale.
Treatment Non-Response Rate | From baseline (Week 1) to post-treatment (Week 10).
  Percentage of eligible patients (i.e., those who start disordered eating treatment) who are deemed as not progressing in therapy as expected (per the CBT-T treatment manual, as determined by the clinician conducting their sessions). To be calculated with the equation: [# of patients who start CBT-T] / [# of patients deemed 'non-responders' by their clinician.]
Treatment Completion Rate | From baseline to 3-month follow-up (i.e., 3 months after Week 10)
  Percentage of eligible patients (i.e., those who start disordered eating treatment) who complete the core treatment (i.e., 10 weekly sessions) and that complete core treatment plus follow-ups (i.e., 1- and 3-month sessions). To be calculated with the equation: [# of patients who start CBT-T] / [# of patients recorded as having completed their prescribed course of treatment by their clinician.]
Program Dropout Rate | From recruitment initiation (Month 0) to recruitment end (Month 24).
  Percentage of eligible patients (i.e., those who initiate the screening procedure) who dropout of the TEAM-ED program.
Acceptability of the TEAM-ED program to clinicians. | At 12 and 18 months.
  Clinicians engaged in the TEAM-ED program will be asked to complete a survey online at ~12 and 18 months into the study (i.e., following the start of recruitment). The objectives of these groups is to: Evaluate the interdisciplinary approach; Identify barriers and facilitators; Assess the perceived effectiveness; and Refine and optimize the model.
Adjunctive Pharmacotherapy Initiation Rate | From baseline to 3-month follow-up.
  Percentage of eligible patients (i.e., those who start disordered eating treatment) who initiate pharmacotherapy for related symptoms during their course of treatment. *This variable is observational - pharmacotherapy initiation is not being directed or controlled by the research protocol or research team.
Patient satisfaction with the TEAM-ED program. | At 3-month follow-up (i.e., 3 months after Week 10).
  Patients in TEAM-ED treatment will participate in a semi-structured, one-on-one interview with a trained research assistant. The objectives of the interviews are to assess overall patient satisfaction with the program including strengths and weaknesses, perceived effectiveness, and areas requiring refinement.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Keshen, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Abbie J Lane Memorial Building, QEII Health Sciences Centre, Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No